CLINICAL TRIAL: NCT00234403
Title: A Phase II Trial to Evaluate the Combination of ZD1839 (Iressa) and Fulvestrant (Faslodex®) in Patients With Advanced or Metastatic Breast Cancer
Brief Title: A Trial to Evaluate the Combination of Iressa & Faslodex® in Patients With Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0141
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: Advanced breast cancer; Metastatic breast cancer; ER positive breast cancer; PR positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib; Fulvestrant

INTERVENTIONS:
Drug: gefitinib and fulvestrant

SUMMARY:
The progression free survival and efficacy of 250 mg ZD1839 in combination with a fixed dose of fulvestrant 250 mg im once a month will be evaluated in female patients with histologically-confirmed advanced or metastatic, ER and/or PR positive breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic breast cancer
* postmenopausal females with amenorrhoea > 12 months and an intact uterus
* FSH levels within postmenopausal range or have undergone a bilateral oophorectomy
* ER &/or PR positive
* previous adjuvant hormone therapy > 12 months prior to enrolment
* previous adjuvant chemotherapy > 6 months prior to enrolment
* measurable disease according to RECIST and/or non measurable bone disease
* life expectancy of at least 12 weeks
* World Health Organisation (WHO) performance status (PS) of 0 to 1.

Exclusion Criteria:

* Male
* life-threatening metastatic visceral disease
* evidence of clinically active interstitial lung disease
* ER and PR negative
* treatment with LHRH analogues < 3 months prior to enrolment
* patients who have restarted menses or do not have FSH levels within the postmenopausal range
* treatment with strontium - 90 (or other radio pharmaceutical) within the previous 3 months
* Treatment with hormonotherapy and/or chemotherapy for advanced disease
* extensive radiotherapy to measurable lesions within the last 4 weeks (i.e. >30% of bone marrow, e.g. whole of pelvis or half of spine)
* currently receiving oestrogen replacement therapy
* treatment with a non-approved or experimental drug within 4 weeks before enrolment
* absolute neutrophil count (ANC) less than 1.5 x 109/litre (L) or platelets less than 100 x 109/L , serum bilirubin greater than 1.25 times the upper limit of reference range (ULRR, serum creatinine greater than 1.5 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULRR if no demonstrable liver metastases, or greater than 5 times the ULRR in the presence of liver metastases, history of bleeding diathesis or long term or present anticoagulant therapy (other than antiplatelet therapy
* any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
* concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, known
* severe hypersensitivity to ZD1839 or fulvestrant or any of the excipients of this product.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-05; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the progression-free survival (PFS) of the combination of 250 mg ZD1839 and fulvestrant in patients with advanced or metastatic breast cancer

SECONDARY OUTCOMES:
To estimate the objective response rate (complete response [CR] and partial response [PR]) at trial closure.
To estimate the disease control rate at trial closure.
To estimate overall survival.
To evaluate the safety & tolerability of the combination gefitinib and fulvestrant

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Spain Medical Director, MD, Study Director — AstraZeneca
Locations (7):
- Spain (7):
  - Investigative Site, Alicante
  - Investigative Site, Girona
  - Investigative Site, Jaén
  - Investigative Site, Madrid
  - Investigative Site, Seville
  - Investigative Site, Valencia
  - Investigative Site, Zaragoza